CLINICAL TRIAL: NCT02158910
Title: A Plan on Investigation and Collection of Aricept Safety Information With a Dose Increase on Alzheimer's Disease Patients
Acronym: AID
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: ART-M082-601
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aricept Group 1: Subjects starting at 5 mg Aricept and increasing their dose to 10 mg Aricept
  Interventions: Drug: Aricept
- Aricept Group 2: Subject starting at 10 mg Aricept and increasing their dose to 23 mg Aricept
  Interventions: Drug: Aricept

INTERVENTIONS:
Drug: Aricept — 5 mg Aricept increasing dose to 10 mg Aricept, or 10 mg Aricept increasing dose to 23 mg Aricept

SUMMARY:
The purpose of the study is for investigation and collection of Aricept safety information with a dose increase on Alzheimer's disease patients.

DETAILED DESCRIPTION:
This is an observational study to systematically investigate domestic patients with Alzheimer's disease to figure out the safety under a situation of the use of Donepezil HCl 23mg. Additionally, if the dose of Donepezil HCl increase, there is need to examine the safety of Donepezil HCl 23mg in depth for patients with Alzheimer's disease by comparing aspects of occurring adverse events by the type of Donepezil HCl increase.

ELIGIBILITY:
Inclusion Criteria

1. Patients who admitted the reading and using of his/her biographical and medical data by word
2. Patients who maintained Aricept dosage for at least 3 months before involved in the study

Exclusion Criteria

1. Hypersensitivity to the active substance or to any of the excipients
2. Breast feeding
3. Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alzheimer's disease
Sampling Method: Non-Probability Sample
Enrollment: 2231 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability due to an increase of Aricept in patients with Alzheimer's disease. | Up to 12 Weeks
  The aspects of adverse events between those who have increased Aricept dosage from 5mg to 10mg and those who have increased Aricept dosage from 10mg to 23mg will be compared. The subjects will be observed at least more than 12 weeks after Aricept administration. The patients who have obtained safety information through a visit after Aricept administration at least once will be selected as the subjects who can be assessed under the status of use.

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Busan
  - Chungcheongbuk-do
  - Chungcheongnam-do
  - Daegu
  - Gangwon-do
  - Gwangju
  - Gyeonggji-do
  - Gyeongsangbuk-do
  - Gyeongsangnam-do
  - Jeju-do
  - Jeollabuk-do
  - Jeollanam-do
  - Seoul